CLINICAL TRIAL: NCT04007146
Title: Systematic Calculation of HyperOxygenation Transit Time Mesure transcutanée de l'oxygène au Cours de l'Hyperoxie Transitoire
Brief Title: Systematic Calculation of HyperOxygenation Transit Time
Acronym: SCHOTT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: With Covid period, inclusions can't be efficient.
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-002571-33
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Output
Keywords: Cardiac Output; vascular medicine; Transcutaneous Oxymetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Output Measurement (Experimental): Subject will have a usual cardiac output
  Interventions: Diagnostic Test: Transcutaneous oxymetry measurement

INTERVENTIONS:
Diagnostic Test: Transcutaneous oxymetry measurement — Transcutaneous oxymetry measurement with transient hyperoxia period (2 periods of 30seconds at 60% of oxygen)

SUMMARY:
Cardiac output (CO) is an essential physiological parameter of healthy person or illness.

In clinical practices, all methods of measuring the CO(Fick method, thoracic impedance, esophageal echodoppler etc) contain limit. Each method are dangerous or hard to implement.

CO is probably determining element of blood transit time and thus the availability of oxygen between the central organs (heart, lung) and the peripheral organs (leg, arms).

Our hypothesis is transcutaneous oxymetry mesurement with oxygen inhalation, to cause a transient hyperoxia, can be used to determinate blood transit time between central organs and peripheral organs. This simple method will be non invasive technique.

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed.

The time of onset hyperoxia will be compare to usual CO method by cross correlation.

The duration of participation for subject is equal to 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* Cardiac output measurement considered at least 2 hours prior to the study
* Affiliation to a French National healthcare system
* Written informed consent must be obtained prior to protocol-specific

Exclusion Criteria:

* Acute or decompensated cardiac or respiratory failure
* Allergy to medical adhesives
* Patients under reinforced protection, pregnancy, deprived of liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social establishment for purposes other than research
* Inability to understand the instructions or objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Estimation of transcutaneous oxymetry with transient hyperoxia | 24 months
  Transition time calcutation from oxygen to peripheral organs by transcutaneous oxymetry method.
Average of CO measured | 24 months
  Average of CO by usual method (catheterisation or transoesophageal echocardiography) reported in medical record of patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MD ABRAHAM, PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: No